CLINICAL TRIAL: NCT07147218
Title: Accelerated Transcranial Magnetic Stimulation for Major Depressive Disorder
Brief Title: Accelerated TMS for MDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-10004-000
Record Dates: First submitted 2025-08-27; First posted 2025-08-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Other): Patients will receive 5 consecutive calendar days of treatments with 6-8 treatments per day for a total of 36 treatments
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — transcranial magnetic stimulation - DASH 36 treatment delivered in 5 days

SUMMARY:
An open-label, multi-center, prospective study to evaluate feasibility and efficacy of accelerated TMS for patients with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
This protocol will investigate the feasibility, tolerability and clinical efficacy of an accelerated TMS protocol delivering 36 sessions in 5 days

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 15 years and older
3. Able to provide informed consent or/and assent
4. Diagnosed with major depressive disorder (MDD) and currently experiencing a major depressive episode (MDE)
5. Adult participants failed to respond to at least one prior anti-depressant medication; for adolescent participants, TMS therapy is used as an adjunct treatment as stated in the FDA cleared indications, but failure to respond adequately to prior anti-depressant medication is not required
6. Participant prescribed TMS Therapy to treat MDD by his or her physician independent of potential participation in this clinical study
7. On a stable antidepressant treatment regimen (whether medication, therapy, other methods or no treatment at all) for at least the past 4 weeks and agrees to remain on the same treatment regimen throughout study enrollment
8. Willing to comply with all the study procedures, complete required assessments and visits, and be available for the duration of the study

Exclusion Criteria:

1. Participants satisfy any one or more of the contraindications for TMS per current treatment guidelines as determined by the PI
2. Total MADRS score of < 20 or PHQ-score <10 at the screen or baseline visits
3. Current diagnosis of substance use disorder (Abuse or Dependence, as defined by DSM-V-TR), with the exception of nicotine dependence
4. Displaying symptoms of substance withdrawal
5. History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes
6. Any disorder which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within six months prior to screening
7. Has a clinically significant abnormality on the screening examination that might affect safety, study participation, or confound interpretation of study results
8. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation
9. History of non-response to TMS or ECT
10. History of any implanted device or psychosurgery for depression
11. PI opinion: Considered at significant risk for suicide during the course of the study
12. Have any medical or psychological condition, that in the opinion of the referring psychiatrist or investigator, would prevent the participant from completing the study, put the participant at unacceptable risk or could interfere with study assessments or integrity of the data

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS score from baseline to post-treatment. | 2 weeks
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-administered tool used to assess the severity of depressive symptoms. Scores range from 0 to 60, with higher scores indicating greater severity

SECONDARY OUTCOMES:
Change in PHQ-9 from baseline to post-treatment. | 2 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a self-report questionnaire used to screen for depression scores range from 0-27 with higher scores indicating greater severity

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Cole, PhD, Study Director — Neuronetics
Locations (3):
- United States (3):
  - Brighter Neurotherapeutics, New York, New York
  - TMS of the Carolinas, Charlotte, North Carolina
  - New chapter TMS, Spokane, Washington